CLINICAL TRIAL: NCT03522831
Title: A Double-blind Placebo-controlled Crossover Study to Assess the Effects of Bronchodilation on Dyspnea, Ventilatory Responses, and Exercise Tolerance in Adults With Cystic Fibrosis
Brief Title: CF Bronchodilation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: H17-02029
Record Dates: First submitted 2018-03-19; First posted 2018-05-11 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Lung Diseases; Cystic Fibrosis
Keywords: dyspnea; exercise endurance; lung disease
MeSH Terms: conditions — Lung Diseases; Cystic Fibrosis; Dyspnea | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol meter-dose inhaler (Active Comparator): Inhalation of 400 μg salbutamol
  Interventions: Drug: Salbutamol
- Placebo meter-dose inhaler (Placebo Comparator): Inhalation of 400 μg placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — Administration of 400 μg meter-dose inhaler of salbutamol performed using large-volume spacer
  Arms: Salbutamol meter-dose inhaler
Drug: Placebo — Administration of 400 μg meter-dose inhaler of placebo performed using large-volume spacer
  Arms: Placebo meter-dose inhaler

SUMMARY:
It is estimated that one in every 3,600 children in Canada has cystic fibrosis (CF). CF is a genetic disease that affects the glands that produce mucus and sweat. In CF, mucus production increases and the mucus becomes thick and sticky. This can block the airways, making it difficult to breathe. Mucus production also causes bacteria to grow, which can lead to infections in the lungs. Individuals with CF suffer from shortness of breath, wheezing, cough, and poor exercise capacity. There are limited treatment options to reduce shortness of breath in these individuals. Some medications known as bronchodilators are commonly prescribed to reduce breathlessness in patients with CF. These drugs help open the airways making it easier to breathe. Unfortunately, there is limited scientific proof that these drugs can reduce shortness of breath and improve exercise capacity in patients with CF. As a result, some experts have recommended that these drugs should not be prescribed for patients with CF. The purpose of this study is to examine the effects of a bronchodilator on shortness of breath, exercise performance, and breathing responses compared to a placebo drug in adults with CF.

DETAILED DESCRIPTION:
BACKGROUND

Exertional dyspnea is a symptom that reduces quality of life and is associated with reduced exercise tolerance in individuals with cystic fibrosis (CF). Lung hyperinflation has been suggested to be an important factor contributing to dyspnea in CF. Dynamic hyperinflation during exercise testing has been reported in up to 58% of CF patients with mild-to-moderate CF lung disease and is associated with reduced exercise tolerance and increased exertional dyspnea.

Dynamic lung hyperinflation also occurs in chronic obstructive pulmonary disease (COPD) and is believed to be a major cause of exertional dyspnea and exercise limitation. Bronchodilator use in COPD has been shown to reduce lung hyperinflation and improve exertional dyspnea and exercise tolerance; however, there is limited data available in CF despite the pathophysiological similarities between these conditions. Although a majority of individuals six years and older with CF are prescribed bronchodilators, evidence to support the chronic use of bronchodilators has been insufficient.

Unlike acute bronchodilator reversibility testing during routine spirometry, cardiopulmonary exercise testing (CPET) is a highly sensitive and reproducible tool to assess the efficacy of bronchodilators in CF. CPET can be used to identify significant physiological abnormalities even in patients with mild CF lung disease with relatively normal spirometry. Compared to healthy age-matched controls during exercise, adults with mild-to-moderate CF have: greater exertional dyspnea; higher ventilatory requirements; earlier constraints on tidal volume expansion; increased operating lung volumes; an earlier onset of unpleasant dyspnea descriptors (i.e. unsatisfied inspiration); and are more likely to experience "chest tightness". All of these abnormalities are, in theory, amenable to change following bronchodilator therapy.

Very few studies have evaluated the effects of short-acting bronchodilators on exercise in CF using CPET. In these studies, despite improvements in forced expiratory volume in one second (FEV1), short-acting β2-agonists (SABA) failed to show any effect on maximal exercise parameters including workload, oxygen uptake, dyspnea, and leg discomfort ratings. Unfortunately, these studies used incremental exercise tests and focused on peak dyspnea responses, which are often unresponsive to most pharmacological and non-pharmacological interventions. A more clinically and physiologically relevant protocol is to use constant work rate exercise tests and to evaluate dyspnea at standardized submaximal exercise times. This approach has been highly effective in showing beneficial effects of bronchodilators in COPD. Accordingly, the purpose of this study is to evaluate the acute effects of SABA on sensory, physiological, and exercise performance outcomes in adults with CF. We hypothesize that SABA will reduce dyspnea intensity ratings and ventilatory limitations, delay the onset of unpleasant dyspnea descriptors, and will improve exercise performance compared to placebo. These findings would support future guideline recommendations for the use of SABAs to improve dyspnea and exercise tolerance in patients with CF.

METHODS

Experimental Overview: This randomized, double-blind, placebo-controlled, crossover study will include a total of four visits to the Cardiopulmonary Exercise Physiology Laboratory at St. Paul's Hospital.

Visit 1 will include medical history screening, chronic activity-related dyspnea, quality of life, and physical activity questionnaires, anthropometric measurements, pulmonary function assessment, and a symptom-limited incremental cycle exercise test to determine peak incremental work rate. On visit 2, participants will perform a constant-load cycle exercise test at 75% of peak incremental work rate (from visit 1) in order to familiarize participants with the exercise protocol and experimental procedures. Visits 3 and 4 will include baseline pulmonary function testing followed by inhalation of either 400 μg salbutamol or matched placebo, in a 2x2 crossover randomized design. Approximately 10 minutes after administration of salbutamol or placebo, subjects will undergo pulmonary function testing and the same constant-load cycle exercise test performed on visit 2. All visits will take place at the same time of day. Visits 1 and 2 will be separated by a minimum of 48 hours and visits 3 and 4 will be separated by a minimum of one week and a maximum of five weeks. Participants will be instructed to perform their usual daily chest physiotherapy and will be required to withhold SABAs, nebulized therapies, and caffeine for a minimum of 6 hours, and long-acting bronchodilators and strenuous exercise for 24 h prior to each visit.

Randomization and Blinding: The random allocation sequence will be computer-generated in blocks of four. Drugs will be prepared as two identical meter-dose inhalers, which will be administered according to the blinded randomization sequence. Drug administration will be performed using identical large-volume spacers. The unblinding code will be held by an individual not involved in the study, and all data collection and analysis will be performed before the treatment codes are broken. All investigators and staff will be unaware of treatment allocations at all times.

Outcome Measures: Primary Efficacy Endpoint: Change in standardized dyspnea score at the highest equivalent submaximal exercise time achieved on both constant load exercise tests (i.e., iso-time) between salbutamol vs. placebo. Secondary Efficacy Endpoints: Exercise endurance time, standardized leg discomfort score, qualitative dyspnea measurements, spirometry, plethysmographic lung volumes, airways resistance, impulse oscillometry derived variables, and metabolic and cardiopulmonary parameters (e.g. ventilatory responses, inspiratory capacity/dynamic hyperinflation, operating lung volumes, expiratory flow limitation, breathing patterns, metabolic responses, and arterial oxygen saturation).

Exercise Protocol: A symptom-limited incremental exercise test will be performed on visit 1 using an electronically braked cycle ergometer (Ergoselect 200P; Ergoline GmbH, Bitz, Germany), according to recommended guidelines for cardiopulmonary exercise testing. The test will consist of steady-state rest for six minutes, a one minute warm-up of unloaded pedaling, and 10-20 watt stepwise increases in work rate, every minute until symptom-limitation using a self-selected cadence. Constant-load exercise tests on visits 2, 3, and 4 will include rest and warm-up periods followed by an immediate increase in work rate to 75% of maximal work (determined on visit 1) until symptom-limitation, using a cadence >50 rpm.

Pulmonary Function: Spirometry, plethysmography, diffusing capacity of the lungs for carbon monoxide, maximum respiratory pressures, and impulse oscillometry will be performed on visit 1, according to established recommendations. Pulmonary function testing on visits 3 and 4 will include spirometry, plethysmography, and impulse oscillometry performed before and ~10 minutes after administration of salbutamol and placebo. A commercially available cardiopulmonary testing system will be used, and all measurements will be expressed as percentage of predicted values.

Dyspnea Evaluation: Dyspnea intensity (defined as "the sensation of laboured or difficult breathing") and perceived leg discomfort will be evaluated at rest, every minute during exercise, and at peak exercise using the modified 0-10 category-ratio Borg scale, on all testing visits. Participants will be asked to select the most applicable dyspnea descriptor(s) after the intensity ratings using the following three descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all three of the descriptors can be chosen at any one time. Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire.

Cardiorespiratory Responses to Exercise: Standard cardio-respiratory measures will be recorded and averaged over 30-second epochs, including minute ventilation, oxygen consumption, carbon dioxide production, tidal volume, and breathing frequency using a commercially available system (Parvo Medics TrueOne 2400). Heart rate will be monitored using a 12-lead electrocardiogram (ECG), blood pressure will be measured using a manual sphygmomanometer, and arterial oxygen saturation will be monitored using pulse oximetry prior to, during, and after all exercise testing.

Operating volumes (i.e., end-expiratory and end-inspiratory lung volumes) will be derived from dynamic inspiratory capacity maneuvers as previously described. Expiratory flow limitation will be measured by placing tidal flow-volume loops within the maximum flow-volume loop. Briefly, a maximum flow-volume loop will be constructed by taking the highest expiratory flows for any given lung volume from a series of graded vital capacity maneuvers performed before and after exercise to account for both thoracic gas compression and exercise-induced bronchodilation. Tidal flow-volume loops will be ensemble averaged and placed within the maximum flow-volume loop according to the measured end-expiratory lung volume. The degree of expiratory flow limitation will be calculated as the percentage overlap between the expired portion of the ensemble averaged tidal flow-volume loop and the maximum flow-volume loop.

Sample Size and Statistical Analyses: The primary endpoint for this study will be dyspnea ratings during exercise at iso-time, defined as the highest equivalent submaximal time achieved during both constant-load exercise tests by a given patient. Using a two-tailed paired subject formula with α=0.05 and β=0.80, we estimate that 16 participants are needed to detect a minimal clinically important difference of ±1 Borg 0-10 scale units at iso-time between treatments, assuming a standard deviation of ±1 Borg 0-10 scale units. Assuming a 20% rate of attrition, at least 20 participants will need to enter the study to ensure adequate power for the primary and secondary endpoints.

Paired t-tests or Wilcoxon signed-rank tests will be used to identify changes in iso-time dyspnea (primary outcome) and secondary outcome measures (e.g. endurance time; iso-time leg discomfort ratings, operating volumes, etc.) comparing salbutamol to placebo. Possible crossover and period effects for all outcomes will be assessed using paired t-tests according to recommended guidelines for design and analysis of crossover trials. Qualitative descriptors of dyspnea and reasons for stopping exercise will be compared using McNemar's test. Multivariate models will be developed to identify predictors of between-test differences in outcomes (e.g. iso-time Borg dyspnea scale and exercise endurance time) for each individual. Predictor variables will include the between-test difference in operating lung volumes, dynamic hyperinflation, and expiratory flow limitation at iso-time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF based on consensus criteria
* Aged 19 years or older
* Stable clinical status
* Pre-bronchodilator FEV1.0 between 30% and 90% predicted
* Body mass index between 16 and 30 kg/m2
* Currently non-smoking or a past smoking history of less than 20 pack-years

Exclusion Criteria:

* A disease other than CF that could importantly contribute to dyspnea or exercise limitation
* Chronic airway infection with Mycobacterium abscessus, Burkholderia cepacia complex, or other organisms with infection control implications according to the treating physicians Contraindications to clinical exercise testing
* Use of supplemental oxygen or desaturation less than 80% with exercise
* History of solid organ transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized dyspnea score at the highest equivalent submaximal exercise time achieved on both constant load exercise tests (i.e., iso-time). | 30 min post-dose.
  Dyspnea rating measured using the Borg 0-10 category ratio scale. Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.

SECONDARY OUTCOMES:
Exercise endurance time on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured during the exercise test following inhalation of drug or placebo.
Ventilatory responses on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Inspiratory capacity/dynamic hyperinflation on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Operating lung volumes on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Expiratory flow limitation on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Breathing patterns on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Metabolic responses on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Arterial oxygen saturation on both constant load exercise tests. | 30 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Standardized leg discomfort score on both constant load exercise tests. | 30 min post-dose.
  Leg discomfort rating measured using the Borg 0-10 category ratio scale. Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Qualitative dyspnea measurements on both constant load exercise tests. | 30 min post-dose.
  Participants will be asked to select the most applicable dyspnea descriptor(s) after the intensity ratings using the following 3 descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all three of the descriptors can be chosen at any one time. Multiple selections are permitted as long as they apply equally. Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason) and to select qualitative descriptors of breathlessness using an established questionnaire. Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest and during the exercise test following inhalation of drug or placebo.
Spirometry on both constant load exercise tests. | 10 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest following inhalation of drug or placebo.
Plethysmographic lung volumes on both constant load exercise tests. | 10 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest following inhalation of drug or placebo.
Airways resistance on both constant load exercise tests. | 10 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest following inhalation of drug or placebo.
Impulse oscillometry on both constant load exercise tests. | 10 min post-dose.
  Parameters will be measured during visits 3 and 4. Each visit is separated by at least one week and a maximum of five weeks. Parameters will be measured at rest following inhalation of drug or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia - Centre for Heart Lung Innovation
Locations (1):
- UBC Cardiopulmonary Exercise Physiology Laboratory, Vancouver, British Columbia, Canada